CLINICAL TRIAL: NCT05847920
Title: A Phase II Seamless Design, Randomized, Double-blind, Placebo-controlled, Dose-exploration Study Evaluate the Efficacy and Safety of SHR-2010 Injection in Patients With Primary IgA Nephropathy
Brief Title: Efficacy and Safety of SHR-2010 Injection in the Treatment of Primary IgA Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the adjustment of the R & D strategy, the sponsor decides to terminate the research.
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2010-201
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2010 Injection (Experimental)
  Interventions: Drug: SHR-2010 Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-2010 Injection — SHR-2010 Injection
  Arms: SHR-2010 Injection
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR - 2010 injection in patients with primary IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Renal biopsy confirmed primary IgA nephropathy
3. 24 hours urinary protein quantity ≥1g, or UPCR≥0.8 g/g
4. eGFR≥30 mL/min/ 1.73m2
5. 40kg≤ Weight ≤100kg
6. Has been treated with optimized supportive treatment. (ACEI or ARB to maximum recommended dose or maximum tolerated dose).

Exclusion Criteria:

1. systemic disease which may cause secondary IgA deposition in the mesangial region
2. Specific type of IgA nephropathy
3. History of severe opportunistic infection
4. A history of chronic or recurrent infection within 1 year prior to screening
5. History of active digestive system within one year
6. Have a malignant tumor or a history of malignant tumor
7. Subjects who have received organ transplants
8. Associated with other serious or poorly controlled systemic diseases
9. Hepatitis, syphilis, human immunodeficiency virus (HIV) infection
10. Received systemic immunosuppressive drugs other than glucocorticoids 8 weeks before screening or during run-in period.
11. Received any systemic glucocorticoid 8 weeks before screening or during run-in period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-06-04 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Part 1: change from baseline in Urine Protein to Creatinine Ratio (UPCR) at 12weeks. | 12 weeks
Part 2: change from baseline in UPCR at 24weeks. | 24 weeks

SECONDARY OUTCOMES:
change from baseline in 24 hours urinary protein at 12 weeks (part 1) | 12 weeks
change from baseline in 24 hours urinary protein at 24 weeks (part 2) | 24 weeks
change from baseline in urinary albumin creatinine ratio (UACR) at 12weeks（Part 1） | 12 weeks
change from baseline in urinary albumin creatinine ratio (UACR) at 24weeks（Part 2）. | 24 weeks
change from baseline in glomerular filtration rate (eGFR) at 12weeks and 24weeks （Part 1）. | 12, 24 weeks
change from baseline in glomerular filtration rate (eGFR) at 24weeks and 36weeks （Part 2）. | 24, 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639